CLINICAL TRIAL: NCT07085013
Title: Effectiveness of Individually Trained Oral Prophylaxis Education on Long-Term Oral Health in Medical and Dental Students: A Two-Year Prospective Cohort Study
Brief Title: Effectiveness of Personalized Oral Hygiene Education in Medical and Dental Students Over Two Years
Acronym: iTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Zvonimir Lukac, Doctor of Dental Medicine, University of Mostar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01-I-1827/21
Record Dates: First submitted 2025-07-14; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Oral Health; Oral Hygiene; Periodontal Health; Dental Plaque; Bleeding on Probing; Health Education
Keywords: iTOP; Oral Health; Oral Hygiene; Dental Plaque; Periodontal Health; Oral Health Education; Preventive Dentistry; Medical Students; Dental Students
MeSH Terms: conditions — Dental Plaque; Health Education

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial using a parallel-group design. Participants were randomly assigned to either an intervention group receiving iTOP oral hygiene training or a control group receiving no training. Both groups were followed over two years with assessments at baseline, 3 months, and 2 years.
Who Masked: Outcomes Assessor
Masking Description: Clinical periodontal assessments were performed by trained examiners who were blinded to the participants' group allocation in order to reduce measurement bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTOP Oral Hygiene Training (Experimental): Participants in this arm received a structured, single-session, small-group training based on the Individually Trained Oral Prophylaxis (iTOP) protocol. The session lasted approximately 45 minutes and was led by certified dental professional. It included personalized assessment, demonstration, and hands-on practice of effective toothbrushing techniques and interdental cleaning. A brief motivational reinforcement session was provided at the 3-month follow-up. Participants received standardized oral hygiene kits at each study visit.
  Interventions: Behavioral: Individually Trained Oral Prophylaxis (iTOP)
- Control - No iTOP Training (No Intervention): Participants in this arm did not receive the iTOP oral hygiene training. They continued their usual oral hygiene routines and received no additional educational interventions. However, they received standardized oral hygiene kits and professional dental cleaning at baseline, 3-month, and 2-year follow-up visits, similar to the intervention group. Clinical assessments were conducted at each time point by blinded examiners.

INTERVENTIONS:
Behavioral: Individually Trained Oral Prophylaxis (iTOP) — The iTOP intervention consists of a single, structured, 45-minute, small-group oral hygiene training session conducted by certified dental professional. The session includes personalized instruction on proper toothbrushing techniques (e.g., Bass technique), use of interdental brushes and floss, and patient motivation. At the 3-month follow-up, participants also received a short reinforcement session. Standardized oral hygiene kits (toothbrush, interdental brushes) were provided at each time point.
  Arms: iTOP Oral Hygiene Training

SUMMARY:
This prospective cohort study is designed to evaluate the long-term effects of individualized oral hygiene education, known as Individually Trained Oral Prophylaxis (iTOP), on oral health outcomes in medical and dental students at the University of Mostar, Bosnia and Herzegovina. Participants will be randomly assigned to either an intervention group receiving personalized oral hygiene training (iTOP) or a control group. Both groups will receive professional dental cleaning and standardized oral hygiene kits. Clinical parameters will be assessed at baseline, after 3 months, and at a 2-year follow-up.

DETAILED DESCRIPTION:
This is a prospective, two-year cohort study conducted at the School of Medicine, University of Mostar (Bosnia and Herzegovina), during the 2021/2022 and 2023/2024 academic years. The study is designed to evaluate the long-term effectiveness of a single-session oral hygiene education program, known as Individually Trained Oral Prophylaxis (iTOP), on periodontal health in medical and dental students.

- Study Population and Setting: Participants include first- and fourth-year students of medicine and dental medicine at the University of Mostar during the 2021/2022 academic year. Eligibility criteria include active enrollment and provision of informed consent. Students with systemic diseases affecting periodontal health (e.g., uncontrolled diabetes) or those using medications known to cause gingival overgrowth will be excluded.

- Study Design: Participants will be randomly assigned using a computer-generated list to either the intervention group (iTOP) or the control group. Group allocation will be concealed from examiners to minimize assessment bias. Both groups will receive professional dental cleaning and standardized oral hygiene kits at each examination point. Clinical assessments will be performed by a board-certified periodontist and a calibrated teaching assistant.

- Intervention: The intervention group will receive individualized oral hygiene instruction based on the certified iTOP methodology. This includes hands-on training in toothbrushing, interdental brush use, and flossing. A follow-up motivational session will be scheduled at 3 months. The control group will receive no structured oral hygiene education beyond standard cleaning and kit distribution. Adherence to oral hygiene recommendations will not be systematically monitored.

- Outcomes and Assessments: The primary clinical outcomes include plaque index, bleeding on probing, probing depth, and clinical attachment level. These will be measured at six sites per tooth using a UNC-15 periodontal probe and recorded on the Bern Periodontal Chart. Assessments are scheduled at baseline (2021/2022), at 3 months, and at the 2-year follow-up (2023/2024). Standardized oral hygiene kits (Curaprox toothbrushes and interdental brushes) will be provided at each time point.

- Statistical Analysis: Planned statistical analyses include both descriptive and inferential methods. Normality will be assessed using the Kolmogorov-Smirnov test. Comparative analyses will use appropriate non-parametric or parametric tests such as the Mann-Whitney U, Wilcoxon signed-rank, Friedman, Chi-square, or Fisher's exact test. All analyses will be conducted using SPSS software (version 26), with significance set at p < 0.05.

- Ethical Considerations: The study was approved by the Ethics Committee of the School of Medicine, University of Mostar (Approval numbers 01-I-1827/21 and 01-I-911/24) and will be conducted in accordance with the Declaration of Helsinki. Written informed consent will be obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Active enrollment as a student in either:
* First or fourth year during the 2021/2022 academic year, or
* Third or sixth year during the 2023/2024 academic year
* Enrollment verified by Faculty Administration records
* Provided written informed consent

Exclusion Criteria:

* Did not provide informed consent
* Presence of systemic conditions known to affect periodontal health (e.g., uncontrolled diabetes, immunodeficiencies)
* Use of medications known to cause gingival overgrowth, including:
* Anticonvulsants
* Calcium channel blockers
* Immunosuppressants

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Change in Plaque Index from Baseline to 2-Year Follow-Up | Baseline, 3 months, and 2 years
  The plaque index was measured using the Bern Periodontal Chart (Periochart) at six sites per tooth, with plaque disclosing agents to identify plaque presence. The outcome is expressed as the percentage of tooth surfaces with visible plaque, ranging from 0% (no plaque present) to 100% (plaque present on all examined surfaces). Higher percentages indicate worse oral hygiene. This measure evaluates the effectiveness of the iTOP intervention in reducing plaque accumulation over time.

SECONDARY OUTCOMES:
Change in Bleeding on Probing from Baseline to 2-Year Follow-Up | Baseline, 3 months, and 2 years
  Bleeding on probing was recorded at six sites per tooth using a UNC-15 probe. This measure evaluates the impact of the iTOP training on gingival inflammation over time.

OTHER OUTCOMES:
Change in Self-Reported Smoking Behavior Over 2 Years | Baseline and 2-Year Follow-Up
  Participants self-reported their smoking status using a study-specific questionnaire administered at baseline and again at the 2-year follow-up. Smoking status was assessed with the question: "Do you currently smoke cigarettes or other tobacco products?", with response options:
  * Yes (current smoker)
  * No (non-smoker)
  Responses were used to calculate the prevalence of smoking within the study population at both time points. The outcome measures the change in smoking behavior over time. Higher prevalence rates reflect greater exposure to a potential confounding factor for periodontal outcomes.
  Note: No standardized or validated scale was used. This was a binary (yes/no) self-report item.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine, University of Mostar, Mostar, HNŽ, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) will be available upon reasonable request to the principal investigator following publication, for research purposes only, and with appropriate data use agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the main results, and will be accessible for up to 5 years.
Access Criteria: Access will be granted to qualified researchers upon reasonable request. Data will include deidentified individual participant data (IPD), study protocol, informed consent form, and statistical analysis plan. Interested researchers should contact the principal investigator via institutional email and provide a brief study proposal and data use agreement.

REFERENCES:
- [Derived] Lukac Z, Maric B, Kapetanovic J, Mandic M, Musa Leko I, Bosnjak AP. Effectiveness of Individually Trained Oral Prophylaxis (iTOP) Education on Long-Term Oral Health in Medical and Dental Students: A Two-Year Prospective Cohort Study. Dent J (Basel). 2025 Sep 3;13(9):404. doi: 10.3390/dj13090404. PMID 41002677